CLINICAL TRIAL: NCT06852638
Title: A Study of the Clinical Application of CD70-targeted PET/ CT Imaging in the Diagnosis of Malignant Cancers
Brief Title: CD70-targeted immunoPET Imaging of Malignant Cancers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LY2024-306-A
Record Dates: First submitted 2025-02-16; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Renal Cancer; Renal Clear Cell Carcinoma; Lymphoma; Lymphoma, Large B-Cell, Diffuse; Follicular Lymphoma; Mantle Cell Lymphoma; Nasopharyngeal Carcinoma
Keywords: The cluster of differentiation (CD70); ImmunoPET; Renal Cancer; Lymphoma; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell; Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD70-targeted immunoPET imaging (Experimental): Enrolled patients will undergo a CD70-targeted immunoPET/CT scanning.
  Interventions: Drug: [18F]F-RESCA-RCCB6; Drug: [18F]F-RESCA-R8B4; Drug: [18F]F-RESCA-RD06; Drug: [68Ga]Ga-NOTA-R8B4; Drug: [68Ga]Ga-NOTA-RD06; Drug: [89Zr]Zr-DFO-RB6; Drug: [89Zr]Zr-DFO-R8B4; Drug: [89Zr]Zr-DFO-RD06

INTERVENTIONS:
Drug: [18F]F-RESCA-RCCB6 — Enrolled patients will receive 0.05-0.1 mCi/kg of [18F]RCCB6. ImmunoPET/CT imaging will be acquired 1-2 hours after [18F]RCCB6 injection.
  Other Names: [18F]RCCB6
Drug: [18F]F-RESCA-R8B4 — Enrolled patients will receive 0.05-0.1 mCi/kg of [18F]R8B4. ImmunoPET/CT imaging will be acquired 1-2 hours after [18F]R8B4 injection.
  Other Names: [18F]R8B4
Drug: [18F]F-RESCA-RD06 — Enrolled patients will receive 0.05-0.1 mCi/kg of [18F]RD06. ImmunoPET/CT imaging will be acquired 1-2 hours after [18F]RD06 injection.
  Other Names: [18F]RD06
Drug: [68Ga]Ga-NOTA-R8B4 — Enrolled patients will receive 0.05-0.1 mCi/kg of [68Ga]R8B4. ImmunoPET/CT imaging will be acquired 1-2 hours after [68Ga]R8B4 injection.
  Other Names: [68Ga]R8B4
Drug: [68Ga]Ga-NOTA-RD06 — Enrolled patients will receive 0.05-0.1 mCi/kg of [68Ga]RD06. ImmunoPET/CT imaging will be acquired 1-2 hours after [68Ga]RD06 injection.
  Other Names: [68Ga]RD06
Drug: [89Zr]Zr-DFO-RB6 — Enrolled patients will receive a single dose (1-3 mCi) of [89Zr]Zr-DFO-RB6 (total 1-2 mg antibody mass). Multiple immunoPET/CT imaging sessions will be performed on day 0, day 1(24 h), day 3 (72 h), day 5 (120 h) or day 7 (168 h).
  Other Names: [89Zr]RB6
Drug: [89Zr]Zr-DFO-R8B4 — Enrolled patients will receive a single dose (1-3 mCi) of [89Zr]Zr-DFO-R8B4 (total 1-2 mg antibody mass). Multiple immunoPET/CT imaging sessions will be performed on day 0, day 1(24 h), day 3 (72 h), day 5 (120 h) or day 7 (168 h).
  Other Names: [89Zr]R8B4
Drug: [89Zr]Zr-DFO-RD06 — Enrolled patients will receive a single dose (1-3 mCi) of [89Zr]Zr-DFO-RD06 (total 1-2 mg antibody mass). Multiple immunoPET/CT imaging sessions will be performed on day 0, day 1(24 h), day 3 (72 h), day 5 (120 h) or day 7 (168 h).
  Other Names: [89Zr]RD06

SUMMARY:
This study aims to establish and optimize the cluster of differentiation (CD70)-targeted immuno-positron emission tomography/computed tomography (immunoPET/CT) imaging method and its physiological and pathological distribution characteristics, based on which the diagnostic efficacy of the above imaging agents in malignant cancers (renal cancer (especially clear cell renal cell carcinoma), lymphoma, or nasopharyngeal carcinoma (NPC)) will be evaluated.

DETAILED DESCRIPTION:
Histologically confirmed malignant cancers (renal cancer (especially clear cell renal cell carcinoma), lymphoma, or nasopharyngeal carcinoma (NPC)), or patients with suspected maligant cancers (renal cancer (especially clear cell renal cell carcinoma), lymphoma, or nasopharyngeal carcinoma (NPC)) indicated by conventional diagnostic imaging will be included. Patients will also be included for routine follow-up, surveillance, and treatment efficacy evaluation.

Enrolled patients will undergo whole-body immunoPET/CT scans 1-2 hours after tracer injection (0.05-0.1 mCi/kg). The uptake of imaging tracers in tumors and normal organs/tissues will be scored visually and quantitatively.

Tumor uptake will be quantified by the maximum standard uptake value (SUVmax). The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and accuracy will be calculated to assess the diagnostic efficacy. The correlation between lesion uptake and CD70 expression level determined by immunohistochemistry staining will be further analyzed. The primary exploration endpoint will be the tracers' imaging feasibility and preliminary diagnostic value compared to conventional imaging approaches like 18F-FDG PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 year-old and of either sex；
* Histologically confirmed diagnosis of renal cancer (especially ccRCC)/lymphoma/NPC or suspected renal cancer/lymphoma/NPC by diagnostic imaging;
* Capable of giving signed informed consent, including compliance with the requirements and restrictions in the informed consent form (ICF) and this protocol.

Exclusion Criteria:

* Pregnancy；
* Severe hepatic and renal insufficiency;
* Allergic to single-domain antibody radiopharmaceuticals.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value (SUV) of normal tissues and organs. | 1 day from injection of the tracers
  Measurement of the overall biodistribution of the above tracers in normal tissues and organs (bladder (after voiding), background (pelvic fat), blood, brain, salivary and lacrimal glands, lung, liver, spleen, pancreas, small intestine, and kidneys). To calculate the SUV, circular regions of interest were drawn around the area of focally increased uptake in the transaxial slices and automatically fitted to a three-dimensional volume of interest.
SUV of tumors | 1 day from injection of the tracers
  The SUV of the above tracers in the primary and/or metastatic lesions of the included subjects. To calculate the SUV, circular regions of interest were drawn around the area of focally increased uptake in the transaxial slices and automatically fitted to a three-dimensional volume of interest.
Radiation dosimetry of tissues/organs | 1 day from injection of the tracers
  Measurement of absorbed radiation doses (Gy/MBq) to tissues/organs. The following tissues were included: adrenals, brain, breasts, gallbladder, small intestine, upper and lower large intestine, stomach, heart contents, heart muscle, kidney, liver, lung, muscle, ovaries, pancreas, red marrow, trabecular and cortical bone, spleen, testes, thymus, thyroid, urinary bladder, and uterus. Dynamic imaging within one hour will be performed for this purpose.
Radiation dosimetry of tumors | 1 day from injection of the tracers
  Measurement of absorbed radiation doses (Gy/MBq) to tumors. Dynamic imaging within one hour will be performed for this purpose.
Radiation dosimetry of whole-body | 1 day from injection of the tracers
  Whole-body activity was measured using a large volume of interest (VOI) covering the entire subject.
Diagnostic sensitivity | 30 days
  Sensitivity = (True Positives) / (True Positives + False Negatives). The diagnostic value of CD70 immunoPET/CT will be compared with that of conventional imaging approaches, including 18F-FDG PET/CT, CT, and MRI.
Diagnostic specificity | 30 days
  Specificity = (True Negatives) / (True Negatives + False Positives). The diagnostic value of CD70 immunoPET/CT will be compared with that of conventional imaging approaches, including 18F-FDG PET/CT, CT, and MRI.
Accuracy | 30 days
  Accuracy = (True Positives + True Negatives) / (Total Tests). The diagnostic value of CD70 immunoPET/CT will be compared with that of conventional imaging approaches, including 18F-FDG PET/CT, CT, and MRI.
Positive Predictive Value (PPV) | 30 days
  PPV = (True Positives) / (True Positives + False Positives). The diagnostic value of CD70 immunoPET/CT will be compared with that of conventional imaging approaches, including 18F-FDG PET/CT, CT, and MRI.
Negative Predictive Value (NPV) | 30 days
  NPV = (True Negatives) / (True Negatives + False Negatives). The diagnostic value of CD70 immunoPET/CT will be compared with that of conventional imaging approaches, including 18F-FDG PET/CT, CT, and MRI.

SECONDARY OUTCOMES:
CD70 immunoPET/CT in altering initial staging for patients with renal cancer/lymphoma/NPC | 3-6 months
  Assess the role of CD70 immunoPET/CT in initial staging in terms of the number of metastases.
CD70 immunoPET/CT for postoperative surveillance for patients with renal cancer/lymphoma/NPC | 3-6 months
  Assess the role of CD70 immunoPET/CT in surveillance in terms of the number of metastases, CD70-derived tumor volume (CD70-TV), and total lesion CD70 uptake (CD70-TLU).
CD70 immunoPET/CT for restaging for patients with renal cancer/lymphoma/NPC | 3-6 months
  Assess the role of CD70 immunoPET/CT in restaging in terms of the number of metastases, CD70-TV, and CD70-TLU.
CD70 immunoPET/CT in evaluating treatment responses | 1-2 years
  We will also investigate the role of CD70 immunoPET/CT in predicting and evaluating the treatment efficacy in patients with renal cancer (especially clear cell renal cell carcinoma, ccRCC), lymphoma, or NPC. The treatment regimens vary for different tumor types but involve chemotherapy, molecularly targeted therapies, immunotherapies (e.g. PD-1/PD-L1 inhibitors), or cell therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Liu, Ph.D. & M.D., Study Chair — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University; Weijun Wei, Ph.D. & M.D., Principal Investigator — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China